CLINICAL TRIAL: NCT01523730
Title: Effects of Repetitive Transcranial Magnetic Stimulation on Cigarette Smoking and Cognitive Function in Smokers With and Without Schizophrenia
Brief Title: Effects of rTMS on Cigarette Smoking and Cognition in Schizophrenia
Acronym: rTMSsmokelab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Tony George, Professor, MD, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: rTMSlab#126/2011
Record Dates: First submitted 2012-01-25; First posted 2012-02-01 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Schizophrenia; Nicotine Addiction
Keywords: Schizophrenia; Nicotine; Transcranial Magnetic Stimulation; Cognition; EEG
MeSH Terms: conditions — Schizophrenia; Tobacco Use Disorder | interventions — Transcranial Magnetic Stimulation; Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Repetitive Transcranial Magnetic Stimulation (rTMS) (Active Comparator)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham rTMS (Placebo Comparator)
  Interventions: Device: Sham Repetitive Transcranial Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Subjects will undergo two testing weeks (active and sham rTMS treatment), washout period ≥ 1 month between the testing weeks. rTMS treatment sessions will take place twice daily on days 1-3 of each test week. Active treatment will be delivered at 90% resting motor threshold intensity. Stimulation will be administered at 20 Hz with 25 stimulation trains of 30 stimuli each with an inter-train interval of 30 sec at equivalent stimulation parameters as those used in our pilot trial. Stimulation Site: Advanced neuronavigation methods will be used to target rTMS to the dorsolateral prefrontal cortex following a T1 weighted MRI scan.
  Other Names: Brain stimulation
  Arms: Repetitive Transcranial Magnetic Stimulation (rTMS)
Device: Sham Repetitive Transcranial Stimulation (rTMS) — Subjects will undergo two testing weeks (active and sham rTMS treatment) administered in a randomized order, to which both experimenter and participant will be blind. There will be a washout period of at least one month between the testing weeks to ensure that any changes in cortical function induced by rTMS have returned to baseline. rTMS treatment sessions will take place twice daily on days 1-3 of each test week. Sham Condition: A single-wing tilt rTMS coil position producing somatic sensation (contraction of scalp muscles) with minimal direct brain effects will be used (same stimulation parameters and site as active condition).
  Arms: Sham rTMS

SUMMARY:
Cigarette smoking rates are extremely high in persons with schizophrenia and this increases the risk of disease and death due to tobacco-related disorders. One of the features of schizophrenia is reduced cognitive abilities, such as poor attention and memory. It is thought that people with schizophrenia smoke cigarettes to reduce these cognitive problems, as nicotine can improve cognitive function in these people. When people with schizophrenia stop smoking it causes further cognitive difficulties, which makes quitting harder for them compared to people without schizophrenia. A method called repetitive transcranial magnetic stimulation (rTMS) allows clinicians to give repeated magnetic pulses through the scalp to cause changes in brain activity and behaviour. rTMS can improve cognitive function in people with schizophrenia. Studies have also shown that rTMS can reduce tobacco craving and consumption of cigarettes. Therefore, we believe that rTMS will improve the cognitive deficits observed during cigarette smoking abstinence and help reduce cravings for cigarettes. Ultimately, rTMS may help smokers with schizophrenia who can't quit smoking with available treatments. This study will examine the effect of rTMS on tobacco cravings and cognitive problems produced by overnight abstinence from cigarette smoking in persons with schizophrenia in comparison to people without mental illness who smoke. Important information about the potential of rTMS for the treatment of cognitive deficits and tobacco addiction in schizophrenia will be obtained. Providing more effective smoking cessation treatments in people with schizophrenia may lead to improved physical and mental health for these patients, who are extremely susceptible to tobacco addiction and tobacco-related illness.

ELIGIBILITY:
Inclusion Criteria for all subjects:

1. Have a Full Scale IQ ≥ 80 as determined by the Shipley-2 which provides an estimate of pre-morbid intelligence
2. Be non-treatment seeking smokers;
3. Have a score greater than 5 on the Fagerstrom Test of Nicotine Dependence (FTND), a 5-item multiple choice questionnaire which assesses nicotine dependence
4. Report smoking of at least 10 cigarettes per day using a self-report 7-day timeline follow-back
5. Have an expired breath CO level >10ppm
6. Be able to provide informed consent.

Inclusion Criteria for Schizophrenia Subjects:

1. Meet SCID for DSM-IV diagnostic criteria for schizophrenia or schizoaffective disorder
2. Be in stable remission from positive symptoms of psychosis as judged by psychiatric evaluation and a PANSS total score <70
3. Be receiving a stable dose of antipsychotic mediation(s) for at least one month.

Inclusion Criteria for Healthy Controls:

1. Do not meet SCID for DSM-IV criteria for any current or past psychiatric disorder except for past major depression if it has been in remission for a minimum of one year
2. Not taking any psychotropic medications

General Exclusion Criteria:

1. Meet criteria for abuse or dependence of alcohol or illicit substances within the past 3 months (with the exception of nicotine dependence or caffeine)
2. Use of nicotine replacement or tobacco products other than cigarettes
3. Concomitant medical illness (including unstable or other presentations thought by investigators to compromise study participation, e.g. diabetes mellitus, hypothyroidism or acute/chronic renal insufficiency) or neurological illness including a history of seizures or a first-degree relative with a history of a seizure disorder
4. Be pregnant or planning to become pregnant
5. Metallic implants.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Cigarette craving as assessed by Tiffany Questionnaire for Smoking Urges (TQSU) | Pre- and post rTMS/sham treatment week 1 and 2: at baseline smoking as usual (day 2), following over-night smoking abstinence (day 3am) and smoking reinstatement (day 3pm)
  Craving will be assessed using the TQSU, a 32-item list of signs and symptoms of nicotine cravings and urges to smoke which subjects rate how strongly they agree or disagree with the statements on a scale of 1 (strongly disagree) to 7 (strongly agree).

SECONDARY OUTCOMES:
Cigarette withdrawal using the Minnesota Nicotine Withdrawal Scale (MNWS) | Pre- and post rTMS/sham treatment week 1 and 2: at baseline smoking as usual (day 2), following over-night smoking abstinence (day 3am) and smoking reinstatement (day 3pm)
  Withdrawal will be assessed using the MNWS on which subjects self-report nicotine withdrawal symptoms including nicotine craving, irritability, anxiety, difficulty concentrating, restlessness, increased appetite or weight gain, depressed mood, and insomnia on a 5-point scale of 1 (none) to 5 (severe). Note: The internal consistencies and test-retest reliability of the MNWS, TQSU and FTND in schizophrenia are comparable to those observed in controls.
Expired breath carbon monoxide (CO) levels | Pre- and post rTMS/sham treatment week 1 and 2: at baseline smoking as usual (day 1 and 2), following over-night smoking abstinence (day 3am) and smoking reinstatement (day 3pm)
  Expired Breath CO (in parts per million; ppm) will be used to biochemically verify smoking status.
Plasma nicotine/cotinine levels | Pre- and post rTMS/sham treatment week 1 and 2: at baseline smoking as usual (day 2), following over-night smoking abstinence (day 3am) and smoking reinstatement (day 3pm)
  Plasma nicotine and cotinine levels will provide and objective measurement of cigarette smoking. Assays will be performed by the CAMH Clinical Laboratory using GC/MS/MS procedures which have been adapted from published procedures.
Continuous Performance Test-X (CPT-X) | Post rTMS/sham treatment week 1 and 2: at baseline smoking as usual (day 2), following over-night smoking abstinence (day 3am) and smoking reinstatement (day 3pm)
  The CPT-X is designed to measure sustained attention and response inhibition. Participants press the space bar as quickly as possible after each letter is presented except when the letter 'X' is presented. Common measures reported include % Hits, % Omissions, % Commissions, Reaction Time, Reactions Time Variability and an Attentional Index (d') Duration: 15 minutes
N-back | Post rTMS/sham treatment week 1 and 2: at baseline smoking as usual (day 2), following over-night smoking abstinence (day 3am) and smoking reinstatement (day 3pm)
  The N-back is designed to measure working memory (WM). This task requires continuous upgrades of the memory store and is suited to studying varying levels of working memory load. Task-load will be parametrically manipulated by varying the interval between targets requiring responses (i.e., 1-back, 3-back) according to previously published methods. The dependent variables of interest will include the average performance and reaction times. Duration:45 minutes.
Spatial Delayed Response (SDR) | Post rTMS/sham treatment week 1 and 2: at baseline smoking as usual (day 2), following over-night smoking abstinence (day 3am) and smoking reinstatement (day 3pm)
  The SDR is designed to measure visuospatial working memory (VSWM). Subjects focus on a central fixation cross on a computer screen. While fixated (staring at the cross), a dot-shaped cue flashes in one of 32 possible locations towards the outer edge of the screen. Then a delay period occurs (5, 15 or 30 seconds). After the delay, the fixation cross returns and the subjects must point on the computer screen where they remember seeing the dot cue. Results are reported as the averaged "distance from target" in cm for the 10 trials at each delay condition. Duration: 15 minutes.
EEG recording during performance of N-back Task | Post rTMS/sham treatment week 1 and 2: at baseline smoking as usual (day 2), following over-night smoking abstinence (day 3am) and smoking reinstatement (day 3pm)
  EEG recording during performance of N-back Task:
  EEG data will be collected using the methods reported in by our lab. A 64-electrode cap and Synamps2 DC-coupled EEG system (Compumedics) will be used. Evoked γ-power from the frontal electrodes will be measured while the participants complete the N-back task.
Hopkins Verbal Learning Test Revised (HVLT-R) | Post rTMS/sham treatment week 1 and 2: at baseline smoking as usual (day 2), following over-night smoking abstinence (day 3am) and smoking reinstatement (day 3pm)
  The HVLT measures verbal learning and memory. The HVLT-R is a verbal list-learning test designed to measure the acquisition of new verbal information using a 12-item word list.Duration: 10 minutes.
Smoking Topography | Week 1 and 2: At baseline, day 2 when smoking as usual and following over-night smoking abstinence day 3
  Smoking patterns will be assessed by measuring aspects of smoking topography (using the CReSS system) such as latency to puff, puff frequency, puff volume, puff duration, inter-puff interval, depth of inhalation and inter-cigarette interval which are postulated to be in vivo measures of smoking reinforcement.The CReSS calculates and stores a number of measures including total number of puffs smoked per session, total puff volume per cigarette, puffs per cigarette, duration of inter-puff interval, average maximum puff velocity, average puff volume and average puff duration.
Spontaneous smoking | Week 1 and 2: Pre- and post rTMS/sham treatment at baseline day 1 and 2 when smoking as usual) and following over-night smoking abstinence day 3
  Spontaneous Smoking will be assessed by self-report using timeline followback (TLFB) methods.

CONTACTS AND LOCATIONS:
Overall Officials: Tony P George, M.D., Principal Investigator — Centre for Addiction and Mental Health, Schizophrenia Program, Toronto, ON, Canada
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research